CLINICAL TRIAL: NCT03530839
Title: Lesser Toe PIP Joint Arthrodesis Versus Resection Arthroplasty: A Randomized Controlled Study
Brief Title: Lesser Toe PIP Joint Arthrodesis Versus Resection Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Principal Investigator, Dr. Ulf Krister Hofmann, Senior physician, University Hospital Tuebingen
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 450/2014BO1
Record Dates: First submitted 2018-04-25; First posted 2018-05-21 (Actual); Last update posted 2018-05-21 (Actual); Status verified 2018-05

CONDITIONS: Claw Toe; Lesser Toe Deformity
Keywords: lesser toe deformity; claw toe; PIP joint; arthrodesis; resection arthroplasty
MeSH Terms: conditions — Hammer Toe Syndrome; Ankylosis | interventions — Arthrodesis

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arthrodesis (Experimental): Arthrodesis of the proximal interphalangeal joint by using a threaded K-wire
  Interventions: Procedure: Arthrodesis
- Resection arthroplasty (Active Comparator): Resection arthroplasty of the proximal interphalangeal joint using a normal K-wire
  Interventions: Procedure: Resection arthroplasty

INTERVENTIONS:
Procedure: Arthrodesis — see study group description
  Arms: Arthrodesis
Procedure: Resection arthroplasty — see study group description
  Arms: Resection arthroplasty

SUMMARY:
Background: The aim of this study was to compare operative outcomes after lesser toe deformity correction with either proximal interphalangeal (PIP) joint arthrodesis or PIP joint resection arthroplasty.

Methods: A prospective randomized controlled trial was performed on 37 patients (48 toes) who underwent one of these two procedures. The Numeric Rating Scale (NRS) for pain, American Orthopaedic Foot and Ankle Society (AOFAS) score, osseous consolidation, and clinical outcome were evaluated preoperatively and at 6 weeks and 6 months postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* Patients with one or more claw toes with rigid PIP joint flexion and extension deformity of the MTP joint scheduled for surgical intervention in the investigator's department

Exclusion Criteria:

* known osteoporosis or other bone metabolism disorders
* prior surgery on the toe scheduled for the intervention
* immunodeficiency or immunosuppressive drug intake
* pregnancy
* non-palpable pulses of the posterior tibial artery or the dorsalis pedis artery
* anticoagulation therapy with the exception of acetylsalicylic acid
* a lack of sufficient physical resilience to allow free self-mobilization and walking.

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Pain | Change from preoperatively to 6 weeks postoperatively and to 6months postoperatively
  Change in pain was evaluated using the Numeric Rating Scale for pain (ranging from 0 (no pain) to 10 (maximum pain))
Function | Change from preoperatively to 6 weeks postoperatively and to 6months postoperatively
  Change in function was evaluated using the American Orthopaedic Foot and Ankle Society score (ranging from 0 (severe impairment) to 100 (no problems with foot))

SECONDARY OUTCOMES:
Osseous consolidation | 6months postoperatively
  Osseous consolidation of the procedure was evaluated using x-rays